CLINICAL TRIAL: NCT03321396
Title: Gut Guarding Gel for Endoscopic Resection to Treat Early Gastroenterological Tumor and Polyps (Evaluation of the Safety of Sodium Alginate Mixed With Calcium Lactate on Endoscopic Mucosal Resection / Endoscopic Submucosal Dissection)
Brief Title: Hydrogel Injection to Assist Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: The Industrial Technology Research Institute (Other); National Cheng Kung University (Other); National Research Program for Biopharmaceuticals, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-106-022
Record Dates: First submitted 2017-09-20; First posted 2017-10-25 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Submucosal Tumor of Gastrointestinal Tract
Keywords: Sodium Alginate; Calcium Lactate; Gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic submucosal dissection (Experimental): All participants in the study received Endoscopic submucosal dissection with Sodium Alginate mixed with Calcium Lactate prior to endoscopic resection.
  Interventions: Device: sodium alginate mixed with calcium lactate

INTERVENTIONS:
Device: sodium alginate mixed with calcium lactate — The product is used in Endoscopic submucosal dissection which is accomplished by steps listed as follows: lesion marking, submucosal injection, mucosal incision, submucosal dissection, then en-bloc resection. It's a new submucosal injection regimen, sodium alginate mixed with calcium lactate, which turned to calcium-alginate gel, we called it as "Gut Guarding Gel".

SUMMARY:
The aim of the investigators' study is to evaluate the mucosa-elevating capacity and clinical safety of Sodium Alginate (SA) mixed with Calcium Lactate in assisting Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection.

DETAILED DESCRIPTION:
The study will evaluate the mucosa-elevating capacity and clinical safety of Gut Guarding Gel (the Sodium Alginate (SA) mixed with Calcium Lactate) in assisting Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection to treat early gastroenterological tumor and polyps.

All participants in the study received Endoscopic submucosal dissection with Sodium Alginate mixed with Calcium Lactate prior to endoscopic resection.

The product is used in Endoscopic submucosal dissection which is accomplished by steps listed as follows: lesion marking, submucosal injection, mucosal incision, submucosal dissection, then en-bloc resection. It's a new submucosal injection regimen, sodium alginate mixed with calcium lactate, which turned to calcium-alginate gel, we called it as "Gut Guarding Gel".

Determine the rates of the delayed bleeding/perforation, postpolypectomy electrocoagulation syndrome, and the late tissue injury.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria in order to be entered into the study:

A. Both genders of patients age 20 or older.

B. Superficial tumors or polyps found either in esophagus, stomach, or large intestine via endoscopic diagnosis.

C. Tumor or polyps ≧ 20 millimeters.

D. Superficial tumor or polyps found either in esophagus, stomach, or large intestine have never received any kind of endoscopic treatment.

E. No evidence of depth of submucosal invasion or metastasis via endoscopy.

Exclusion Criteria:

If patients meet any of the following criteria they may not be entered into the study:

A. Patients suffering from other advanced malignant tumors.

B. White Blood Cell< 2000 μL or Severe thrombocytopenia（Platelet count < 50,000 μL)，or blood coagulation abnormalities uncorrectable .

C. Patients taking anti- thrombocytopenia or anti-coagulation medicine, and medication cannot be stopped under physicians' consideration.

D. Main organs (heart, lung, liver, kidney) dysfunction who are not eligible for clinical trials under physicians' consideration.

E. Evidence of depth of submucosal invasion or metastasis via endoscopy.

F. Unable to follow-up by endoscopy.

G. Unwilling to sign informed consent.

H. Allergic to pharmaceutical excipients related to this medical device (Calcium Lactate or Sodium Alginate).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jui-Wen Kang, Study Director — Department of Internal Medicine, National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusano T, Etoh T, Akagi T, Ueda Y, Shiroshita H, Yasuda K, Satoh M, Inomata M, Shiraishi N, Kitano S. Evaluation of 0.6% sodium alginate as a submucosal injection material in endoscopic submucosal dissection for early gastric cancer. Dig Endosc. 2014 Sep;26(5):638-45. doi: 10.1111/den.12268. Epub 2014 Mar 24. PMID 24655031
- [Background] Norouzi M, Nazari B, Miller DW. Injectable hydrogel-based drug delivery systems for local cancer therapy. Drug Discov Today. 2016 Nov;21(11):1835-1849. doi: 10.1016/j.drudis.2016.07.006. Epub 2016 Jul 14. PMID 27423369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started in January 2017. The location was taken place at National Cheng Kung University Hospital. Patients who met the inclusion criteria were recruited.
Period: Overall Study
Arm/Group | Endoscopic Submucosal Dissection
Started | 13
Completed | 12
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Endoscopic Submucosal Dissection
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Postpolypectomy Electrocoagulation Syndrome
Description: To evaluate patient's clinical symptoms and patient's complaints about the post-polypectomy electrocoagulation syndrome. The post-polypectomy electrocoagulation syndrome occurs after performing the endoscopy, and its signs and symptoms are similar to the signs and symptoms of perforation, such as severe abdominal pain and fever.
Time Frame: 5 days after resection
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Submucosal Dissection
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Number of Patients With Delayed Bleeding/Perforation
Description: Perform the endoscopy to evaluate the delayed of bleeding/perforation after 4 weeks of hydrogel injection.
Time Frame: An average of 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Submucosal Dissection
Number analyzed (Participants) | 12
Participants | 1

3. Secondary Outcome: Number of Patients With Late Tissue Injury
Description: To keep follow up the patient's clinical symptoms to evaluate the delayed of bleeding/perforation after one month of hydrogel injection.
Time Frame: One month after endoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Submucosal Dissection
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 weeks.
Description: No adverse events occurred, such as fever, severe abdominal pain and delay-bleeding.
Arm/Group | Endoscopic Submucosal Dissection
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endoscopic Submucosal Dissection (N=12)
Intraprocedural perforation (Gastrointestinal disorders) | 1 (1)
Intraprocedural bleeding (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Only 12 patients completed the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03321396/Prot_SAP_001.pdf